CLINICAL TRIAL: NCT06321874
Title: Exploring Postoperative Effects of Hyperoxic Intermittent Stimuli on Reticulocytes Levels in Abdominal Surgery: A Randomized Single-blind Study
Brief Title: Effects of Oxygen After Abdominal Oncological Surgery
Acronym: EPHIRAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EPHIRAS
Record Dates: First submitted 2024-02-22; First posted 2024-03-20 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-02

CONDITIONS: Abdominal Cancer
Keywords: oncology; abdominal surgery; oxygen
MeSH Terms: conditions — Neoplasms | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: Randomization was conducted post-surgery in a 1:1 ratio across groups: Normobaric Oxygen Paradox (NOP) group, and a control (CTR) group. The NOP group received 60% oxygen for two hours on days 1, 3, and 5 post-surgery using a venti-mask. The CTR group did not receive oxygen therapy during the post-operatory period starting from day 1. All patients could receive oxygen during the surgery and the first 24 hours post-surgery (day 0) as needed. The belonging to one group or the other was blinded to the laboratory staff.
Who Masked: Care Provider
Masking Description: The belonging to one group or the other was blinded to the laboratory staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normobaric Oxygen Paradox (NOP) group (Experimental): The NOP group received 60% oxygen for two hours on days 1, 3, and 5 post-surgery using a venti-mask.
  Interventions: Procedure: Oxygen
- Control (CTR) group (No Intervention): The CTR group did not receive oxygen therapy during the post-operatory period starting from day 1.

INTERVENTIONS:
Procedure: Oxygen
  Arms: Normobaric Oxygen Paradox (NOP) group

SUMMARY:
The aims of the research is to determine whether a Hyperoxic intermittent stimuli protocol can increase reticulocyte counts, signififying a rise in EPO production, in patients undergoing abdominal surgery

DETAILED DESCRIPTION:
For anemia treatment in cancer patients, human recombinant erythropoietin is often used. However, its application is constrained due to high costs, side effects, and limited availability in some regions. This research and clinical exploration aim to identify an tool alternative to transfusion.

Randomization was conducted post-surgery in a 1:1 ratio across groups: Normobaric Oxygen Paradox (NOP) group, and a control (CTR) group. The NOP group received 60% oxygen for two hours on days 1, 3, and 5 post-surgery using a venti-mask. The CTR group did not receive oxygen therapy during the post-operatory period starting from day 1. All patients could receive oxygen during the surgery and the first 24 hours post-surgery (day 0) as needed. The belonging to one group or the other was blinded to the laboratory staff.

Pre-surgery, all patients were administered an oral benzodiazepine. General anesthesia was employed, potentially combined with epidural techniques and standard anesthesia monitors were used. The choice of anesthesia technique was at the discretion of the anesthetist. During surgery, patients received 40-50% FiO2 ventilation and were extubated at the surgery's end. Post-surgery, patients were admitted to the ICU for at least 24 hours, receiving oxygen if saturation dropped below 98%. The oxygen protocol commenced 24 hours after ICU admission (day 1). The transfusion threshold was set at 8 g/dl with clinical signs.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing abdominal oncological surgery

Exclusion Criteria:

* GFR<60 ml/minute and/ or creatinine serum level > 2mg/dl
* Transfusion of red blood cells per or postoperatively
* Bleeding requiring repeated transfusions during or after surgery
* Severe respiratory syndrome necessitating continuous oxygen
* Intolerance to oxygen mask

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2011-11-01 (Actual); Study Completion 2011-11-01 (Actual)

PRIMARY OUTCOMES:
Percentage change in reticulocyte count | 6 days
  Percentage change in reticulocyte count from baseline to day six within each group

SECONDARY OUTCOMES:
haematocrit levels mesure | 6 days
  haematocrit levels mesured at baseline and on day six
haemoglobin levels mesure | 6 days
  haemoglobin levels mesured at baseline and on day six

CONTACTS AND LOCATIONS:
Overall Officials: Maher Khalife, MD, Principal Investigator — Jules Bordet Institute
Locations (1):
- Khalife Maher, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No